CLINICAL TRIAL: NCT06300359
Title: Prognostic Indicators of Gullian-Barre Syndrome at Assiut University Children Hospital
Brief Title: Prognostic Indicators of Gullian-Barre Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Abdelhakem Sayed Amin, Pricipal Investigator, Assiut University
Other Study IDs: Prognostic indicators of GBS
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Guillain-Barre Syndrome
Keywords: Prognostic indicators
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prognostic indicators of Gullian-Barre syndrome and the predictive factors associated with worse prognosis in the Guillain-Barré syndrome (GBS), which can be helpful to fully evaluate the disease progression and provide proper treatments.

DETAILED DESCRIPTION:
Guillain Barre Syndrome (GBS) is an autoimmune disorder with post-infectious polyneuropathy involving motor, sensory and sometimes the autonomic nerves. With the eradication of wild polio virus infection, GBS has become the most common cause of acute flaccid paralysis in both the developed and developing countries.GBS occurs throughout the world with a median annual incidence of 1.3 cases per population of 100 000.

GBS is characterized by ascending paralysis (lower limb numbness, paraesthesia or pain followed by weakness which ascends symmetrically and gradually progresses over a period of 1 to 28 days with maximum severity of weakness by four weeks after the onset). Bulbar involvement is seen in 50% cases and autonomic disturbances are seen in about 20%. Since there may be mortality related to acute complications of respiratory muscle paralysis and morbidity related to the long duration of the paralysis.

It can be classified electrophysiologically into demyelinating and axonal subtypes. Acute inflammatory demyelinating polyneuropathy (AIDP) is the demyelinating subtype, while acute motor axonal (AMAN) and acute motor-sensory axonal neuropathy (AMSAN) are the axonal subtypes. It is difficult to differentiate between them clinically and nerve conduction studies (NCS) can play an important role. Determining the electrophysiological subtype is useful as it can give insights into the underlying pathophysiology. This has both therapeutic and prognostic significance. Various electrodiagnostic criteria sets have been proposed to differentiate between the demyelinating and axonal subtypes.

GBS typically occurs after an infectious disease (Two-thirds of patients report symptoms of a respiratory or gastrointestinal tract infection before the onset of GBS. In about half of patients with GBS, a specific type of preceding infection can be identified and Campylobacter jejuni is responsible for at least one-third of these infections. Other pathogens that cause antecedent infections related to GBS are cytomegalovirus, Epstein- Barr virus, Mycoplasma pneumonia, Haemophilus influenzae, and influenza A virus) in which the immune response generates antibodies that crossreact with gangliosides at nerve membranes. This autoimmune response results in nerve damage or functional blockade of nerve conduction. The type of preceding infection and the specificity of the antiganglioside antibodies largely determine the subtype and clinical course of GBS.

The chance of recovery was significantly affected by age, antecedent gastroenteritis, disability, electrophysiological signs of axonopathy, latency to nadir and duration of active disease.The main treatments did not seem to affect the chance of recovery.

Acute motor axon neuropathy, diabetes, high blood pressure, uroschesis, high body temperature, ventilator support,consciousness disorder, absence of upper respiratory tract preceding infection, hyperglycemia, hyponatremia,hypoalbuminemia, high leukocyte count, hyperfibrinogenemia, abnormal hepatic and renal function were demonstrated as poor prognostic factors.

Dysautonomic syndrome, cardiac arrest and respiratory failure were the leading causes of death.

Paralysis of respiratory muscles is a dreaded complication that occurs in one-fourth of the subjects. Respiratory weakness occurs due to the involvement of both inspiratory and expiratory muscles. Diaphragmatic weakness occurs due to phrenic nerve demyelination. Careful and close monitoring is mandatory to identify patients at high risk for respiratory failure, and triage them to the Intensive Care Unit (ICU) and mechanical ventilation.

The diagnosis was based mostly on clinical judgement and was confirmed by autopsy only in a few instances. In the presence of suggestive findings the complementary test as demyelinising changes in the nerve conduction studies (NCS) or albuminocytological dissociation in the cerebrospinal fluid (CSF), help to confirm the diagnosis.

* Consider specific treatment with IVIg or PE:

  * IVIg is usually the first- line therapy for children with GBS. Although some paediatric centres administer IVIg as 2 g/kg (body weight) over 2 days, rather than the standard adult regimen of 2 g/kg (body weight) over 5 days.
  * plasma exchange can be difficult to perform in young children, and care should be taken in patients with autonomic cardiovascular instability because of the large volume shifts involved in the plasma exchange procedure.

    1. Indications to start IVIg or PE:

       Severely affected patients (inability to walk unaided, GBS disability scale ≥3).

       Unknown whether IVIg is effective:

       Mildly affected patients (GBS disability scale ≤2) or MFS patients .
    2. Indications for re-treatment with IVIg:
  * Secondary deterioration after initial improvement or stabilisation (treatment-related fluctuation): treat with 0·4 g/kg for 5 days.
  * No proven effect of re-treatment with IVIg in patients who continue to worsen.
* Steroids :

Oral steroids or intravenous methylprednisolone (500 mg daily for 5 consecutive days) alone are not beneficial in GBS. The combination of IVIg and intravenous methylprednisolone was not more effective than IVIg alone.

-Give good general care: Monitor progression and prevent and manage potentially fatal complications.

* Indication for admission to an intensive care unit:

  * Rapid progressive severe weakness often with impaired respiration (vital capacity <20 mL/kg).
  * Need for artifi cial ventilation Insufficient.
  * swallowing with high chance of pulmonary infection.
  * Severe autonomic dysfunction.
* Physiotherapy and Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 - 18 years old with guillian barrie syndrome admitted at Assiut university children hospital.

Acceptance to participate in this study .

Exclusion Criteria:

* Patients aged less than 2 years and more than 18 years old . Children or Parents who refused to participate in this study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with GBS, presenting with weakness, diagnosed on clinical and/or electrophysiological grounds, were enrolled. The enrolled children underwent a detailed clinical-assessment followed by nerve conduction studies.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Prognostic indicators of Gullian-Barre syndrome | Baseline
  The predictive factors with worse prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Sayed Amin, Resident, Principal Investigator — Assiut University; Gamal A Abdelaal Asker, Professor, Study Director — Assiut University; Azhar A Mohammed Mohammed, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Berg B, Walgaard C, Drenthen J, Fokke C, Jacobs BC, van Doorn PA. Guillain-Barre syndrome: pathogenesis, diagnosis, treatment and prognosis. Nat Rev Neurol. 2014 Aug;10(8):469-82. doi: 10.1038/nrneurol.2014.121. Epub 2014 Jul 15. PMID 25023340
- [Background] The prognosis and main prognostic indicators of Guillain-Barre syndrome. A multicentre prospective study of 297 patients. The Italian Guillain-Barre Study Group. Brain. 1996 Dec;119 ( Pt 6):2053-61. PMID 9010009
- [Background] van Doorn PA, Ruts L, Jacobs BC. Clinical features, pathogenesis, and treatment of Guillain-Barre syndrome. Lancet Neurol. 2008 Oct;7(10):939-50. doi: 10.1016/S1474-4422(08)70215-1. PMID 18848313
- [Background] Gonzalez-Suarez I, Sanz-Gallego I, Rodriguez de Rivera FJ, Arpa J. Guillain-Barre syndrome: natural history and prognostic factors: a retrospective review of 106 cases. BMC Neurol. 2013 Jul 22;13:95. doi: 10.1186/1471-2377-13-95. PMID 23876199
- [Background] Kuwabara S. Guillain-Barre syndrome: epidemiology, pathophysiology and management. Drugs. 2004;64(6):597-610. doi: 10.2165/00003495-200464060-00003. PMID 15018590
- [Background] Leonhard SE, Mandarakas MR, Gondim FAA, Bateman K, Ferreira MLB, Cornblath DR, van Doorn PA, Dourado ME, Hughes RAC, Islam B, Kusunoki S, Pardo CA, Reisin R, Sejvar JJ, Shahrizaila N, Soares C, Umapathi T, Wang Y, Yiu EM, Willison HJ, Jacobs BC. Diagnosis and management of Guillain-Barre syndrome in ten steps. Nat Rev Neurol. 2019 Nov;15(11):671-683. doi: 10.1038/s41582-019-0250-9. Epub 2019 Sep 20. PMID 31541214
- [Background] Mani AM, Prabhakar AT, Alexander PT, Nair A, Vijayaraghavan A, Shaikh A, Benjamin R, Sivadasan A, Mathew V, Aaron S, Alexander M. Utility of Serial Nerve Conduction Studies in the Electrodiagnosis of Guillain-Barre Syndrome. Neurol India. 2021 Mar-Apr;69(2):369-375. doi: 10.4103/0028-3886.314529. PMID 33904455
- [Background] Nagappa M, Netto AB, Taly AB, Kulkarni GB, Umamaheshwara Rao GS, Periyavan S, Rao S. Electrophysiological observations in critically ill Guillain-Barre syndrome. Neurol India. 2016 Sep-Oct;64(5):914-20. doi: 10.4103/0028-3886.190271. PMID 27625229
- [Background] Rangan RS, Tullu MS, Deshmukh CT, Mondkar SA, Agrawal M. Clinical Profile and Outcome of Guillain-Barre Syndrome in Pediatric Patients Admitted to a Tertiary Care Centre: A Retrospective Study. Neurol India. 2021 Jan-Feb;69(1):81-84. doi: 10.4103/0028-3886.310112. PMID 33642275
- [Background] Zhang Y, Zhao Y, Wang Y. Prognostic factors of Guillain-Barre syndrome: a 111-case retrospective review. Chin Neurosurg J. 2018 Jun 18;4:14. doi: 10.1186/s41016-018-0122-y. eCollection 2018. PMID 32922875
- [Background] Kleyweg RP, van der Meche FG, Schmitz PI. Interobserver agreement in the assessment of muscle strength and functional abilities in Guillain-Barre syndrome. Muscle Nerve. 1991 Nov;14(11):1103-9. doi: 10.1002/mus.880141111. PMID 1745285
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475